CLINICAL TRIAL: NCT04205409
Title: Nivolumab for Relapsed or Refractory Disease Post Chimeric Antigen Receptor T-Cell Treatment in Patients With Hematologic Malignancies
Brief Title: Nivolumab for Relapsed, Refractory, or Detectable Disease Post Chimeric Antigen Receptor T-cell Treatment in Patients With Hematologic Malignancies
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Rahul Banerjee, MD, Assistant Professor, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1005491; NCI-2019-08192 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10388 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2019-12-17; First posted 2019-12-19 (Actual); Results first posted 2025-11-03 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Recurrent Chronic Lymphocytic Leukemia; Recurrent Diffuse Large B-Cell Lymphoma; Recurrent Follicular Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Grade 3a Follicular Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Non-Hodgkin Lymphoma; Recurrent Plasma Cell Myeloma; Refractory Chronic Lymphocytic Leukemia; Refractory Diffuse Large B-Cell Lymphoma; Refractory Follicular Lymphoma; Refractory Marginal Zone Lymphoma; Refractory Non-Hodgkin Lymphoma; Refractory Plasma Cell Myeloma; Recurrent Mantle Cell Lymphoma; Refractory Mantle Cell Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Non-Hodgkin; Multiple Myeloma; Lymphoma, Mantle-Cell | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (nivolumab) (Experimental): Patients receive nivolumab IV over 30 minutes on day 1. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Nivolumab

INTERVENTIONS:
Biological: Nivolumab — Given IV
  Other Names: 946414-94-4; BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo; CMAB819; Nivolumab Biosimilar CMAB819

SUMMARY:
This phase II trial studies how well nivolumab works for the treatment of hematological malignancies that have come back (relapsed), does not respond (refractory), or is detectable after CAR T cell therapy. Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
OUTLINE:

Patients receive nivolumab intravenously (IV) over 30 minutes on day 1. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days and then for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of the following tumor types

  * Non Hodgkin-lymphoma, including:

    * Diffuse large B-cell lymphoma: Histopathologic confirmation
    * Mantle cell lymphoma: Histopathologic confirmation
    * Follicular lymphoma, all grades: Histopathologic confirmation
    * Marginal zone lymphoma: Histopathologic confirmation
  * Chronic lymphocytic leukemia: Histopathologic or flow cytometric confirmation
  * Multiple myeloma: Histopathologic or flow confirmation
* Relapsed, refractory, or detectable disease after treatment with chimeric antigen receptor T-cells

  * Multiple Myeloma: patients must have exhausted all treatment options known to provide clinical benefit, and are refractory to a minimum of 3 prior lines of therapy (including an immunomodulatory imide drug [IMiD], proteasome inhibitor [PI], or anti-CD38 monoclonal antibody)
* Have measurable disease, defined by histology:

  * Non-Hodgkin's lymphoma, based on presence of lesions >= 1.5 cm that can be accurately measured in 2 dimensions by computed tomography (CT) (preferred) or magnetic resonance imaging (MRI), and are not included in any prior field of radiation therapy
  * Chronic lymphocytic leukemia: circulating lymphocytes >= 5,000 / mm^3
  * Multiple myeloma, based on the International Myeloma Working Group (IMWG) criteria of having one or more of the following findings:

    * Serum M protein >= 1.0 g/dL
    * Urine M protein >= 200 mg/24 hours
    * Involved serum free light chain level >= 10 mg/dL with abnormal kappa/lambda ratio
    * Measurable biopsy-proven plasmacytomas (>= 1 lesion has a single diameter >= 2 cm)
    * Bone marrow plasma cells >= 30%
* Age 18 years and older, and have the capacity to give informed consent
* Anticipated survival of > 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Post CAR T cell receipt of intervening palliative radiation therapy is allowed
* Estimated glomerular filtration rate (eGFR) >= 20 ml/min
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 x upper limit of normal (ULN)
* Total bilirubin =< 2 x ULN
* Absolute neutrophil count (ANC) >= 1,000/uL
* Platelets >= 50,000/uL
* Hemoglobin >= 8 g/dL

Exclusion Criteria:

* Receipt of intervening therapy after CAR T-cell infusion
* History of another primary malignancy that has not been in remission for at least 1 year (with the exception of non-melanoma skin cancer, curatively treated localized prostate cancer, curatively treated superficial bladder cancer and cervical carcinoma in site on biopsy or a squamous intraepithelial lesion on papanicolaou [PAP] smear)
* Active hepatitis B, hepatitis C at time of screening
* Known (human immunodeficiency virus [HIV]) seropositivity
* Subjects with uncontrolled infection
* Concurrent use of other anticancer agents or experimental treatments
* Active autoimmune disease requiring immunosuppressive therapy with the exception of vitiligo and autoimmune alopecia
* Known active central nervous system (CNS) involvement
* Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids, and adrenal replacement doses are permitted in absence of active autoimmune disease
* Known history of any active infectious pneumonitis
* Presence of acute or chronic graft-versus-host disease (GVHD) requiring active treatment unless limited to skin involvement and managed with topical steroid therapy alone
* Has active cytokine release syndrome
* Pregnancy or breastfeeding: Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (urine pregnancy test: minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [hCG]) within 14 days of the first dose of study drug. Women must not be breastfeeding. Females of non-childbearing potential are those who are postmenopausal greater than 1 year or who have had a bilateral tubal ligation or hysterectomy. Females of childbearing potential and males who have partners of childbearing potential must agree to use 2 effective contraceptive methods during the study and for 8 months following the last dose of nivolumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-06-05 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2029-08-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Banerjee, MD, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (nivolumab)
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (nivolumab)
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 8
Age, Continuous [Mean (Full Range); unit: years] | 61 [40 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 17
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response Rate (ORR)
Description: Assessed by disease-specific guidelines: multiple myeloma - International Myeloma Working Group response criteria, non-Hodgkin lymphoma - Response assessment will be based on the Lugano Criteria, and chronic lymphocytic leukemia - Response assessment based on the International Workshop on Chronic Lymphocytic Leukemia (IWCLL) Criteria. ORR will be estimated, and its corresponding 95% exact binomial confidence interval (CI) will be provided.
Time Frame: Up to 1 year 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (nivolumab)
Number analyzed (Participants) | 20
Participants | 2

2. Secondary Outcome: Overall Survival
Description: Will employ Kaplan-Meier and Cox proportional hazard model methodology.
Time Frame: From the first study drug administration to death from any cause, up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (nivolumab)
Number analyzed (Participants) | 20
Participants | 8

3. Secondary Outcome: Progression-free Survival
Description: Will employ Kaplan-Meier and Cox proportional hazard model methodology.
Time Frame: From first study drug administration to the first occurrence of disease progression or death from any cause, assessed up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (nivolumab)
Number analyzed (Participants) | 20
Participants | 0

4. Secondary Outcome: Duration of Response
Description: Will employ Kaplan-Meier and Cox proportional hazard model methodology.
Time Frame: Up to 5 years
Reporting Status: Not Posted

5. Secondary Outcome: Incidence of Adverse Events
Description: Will be determined by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0. Safety data will be summarized descriptively. Adverse events will be summarized by severity, seriousness, and relationship to study drug.
Time Frame: Up to 30 days after the last dose of study drug, up to a maximum of 1 year 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (nivolumab)
Number analyzed (Participants) | 20
Participants | 20

ADVERSE EVENTS:
Time Frame: Adverse events are collected from time of consent through 30 days after last dose of study drug, up to a maximum of 1 year 9 months. Deaths were assessed for up to 5 years.
Arm/Group | Treatment (nivolumab)
All-Cause Mortality (participants affected / at risk) | 12/20
Serious Adverse Events (participants affected / at risk) | 10/20
Other Adverse Events (participants affected / at risk) | 18/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (nivolumab) (N=20)
Atrial fibrillation with RVR (Cardiac disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Cardiac arrest (Cardiac disorders) | 1 (1)
Chest pain (Cardiac disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Disease progression (General disorders) | 1 (1)
Febrile neutropenia (General disorders) | 2 (3)
Fever (General disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Lung infection (Infections and infestations) | 1 (1)
Pneumonitis (Infections and infestations) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 3 (5)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (nivolumab) (N=20)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 2 (2)
Blurred vision (Eye disorders) | 1 (1)
Body aches (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 5 (6)
Dizziness (Nervous system disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fatigue (General disorders) | 6 (6)
Fecal incontinence (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Flu like symptoms (General disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Gas (Gastrointestinal disorders) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (3)
Hypertension (Vascular disorders) | 1 (4)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 5 (6)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 6 (10)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Fragility (Skin and subcutaneous tissue disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Peripheral neuropathy (Nervous system disorders) | 1 (1)
Platelet count decreased (Investigations) | 4 (8)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural infection (Infections and infestations) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2)
Small intestinal bacterial overgrowth (Gastrointestinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Steatorrhea (Gastrointestinal disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Watering eyes (Eye disorders) | 1 (1)
White blood cell decreased (Investigations) | 4 (4)
Jaw pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Vision decreased (Eye disorders) | 1 (1)
Pharyngeal congestoin (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-16): https://cdn.clinicaltrials.gov/large-docs/09/NCT04205409/Prot_SAP_001.pdf
  • Informed Consent Form (2021-10-04): https://cdn.clinicaltrials.gov/large-docs/09/NCT04205409/ICF_000.pdf